CLINICAL TRIAL: NCT02762695
Title: Evaluation of a Model of Care for People With Hypertension and Type II Diabetes Based on Case Management and Risk Adjustment
Brief Title: Effectiveness of a Case Management Model for Patients With Hypertension and Type II Diabetes in Chile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Fernando Poblete Arrué, MD, MPH, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-277; ID15I10277 (Other Grant/Funding Number: FONDEF/CONICYT)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
Keywords: Hypertension; Diabetes Mellitus, Type 2; Case Management
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case Management (Experimental)
  Interventions: Other: Case Management
- Control (Active Comparator): Usual Care at Primary Health Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Case Management — A model of health care for chronic patients, based on Case Management and guided by a nurse which targets the patient´s risk.
  The core elements of this strategy are: a. processes to identify specific population and their risk; b. evidence-based practice guidelines according to risk (higher risk, more interventions and monitoring by a nurse, lower risk, higher emphasis on self-care); c. Practice models based on collaboration between health team members leaded by a nurse; d. self-management education for patients; e. monitoring patients face to face or by telephone to ensure to follow the care program (blood test, medical consultation, for example); e. measurement of process and outcomes.
  Arms: Case Management
Other: Usual Care — Usual Care at Primary Health Care Center
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate whether a new model of health care for chronic patients, based on Case Management and guided by a nurse which targets the patient´s risk, is more effective than usual care at Primary Health care in Chile. Additionally, this intervention would provide a better quality of care and a more efficient health provision.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with Hypertension and/ or Type 2 Diabetes

Exclusion Criteria:

* Severe mental illness and / or deterioration of cognitive abilities.
* Severe hearing loss.
* Diagnosed with cancer
* Stage 4 or 5 of chronic kidney disease

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2016-05-04 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin | One year
Systolic and Diastolic Blood Pressure | One year

SECONDARY OUTCOMES:
Quality of Care | one year
  Measured by Clinical records audits
Patient satisfaction | one year
  Measured by a questionnaire
Medication adherence | one year
  Measured by Morisky- Green questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C Poblete, Master, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- CESFAM La Faena, Peñalolén, RM, Chile

IPD SHARING:
Plan to Share IPD: No